CLINICAL TRIAL: NCT04761445
Title: Comparison Between Two Different Tissue-Level Implant Systems: A Prospective Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Sandrine Abi Rached, Principal Investigator, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMD187
Record Dates: First submitted 2020-12-16; First posted 2021-02-21 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Peri-implant Bone Loss; Implant Stability; Vertical Soft Tissue Thickness
Keywords: Marginal bone loss; Crestal bone stability
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Intervention Model Description: The study is designed as a prospective clinical trial with a parallel design comparing two different tissue-level implants placed adjacently in the posterior maxilla and mandible.
Who Masked: Participant
Masking Description: The day of the surgery, each implantation site was given a number depending on the tooth missing. Then, using a random team generator software (Keamk) each site was randomly assigned to one of the two groups based on the implant system used.
  Participants were blinded as to the assignment in the first or second group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Straumann Standard Plus (SP) (Experimental): Patients receiving Straumann SP implants of 4.1 mm in diameter and length of 10 mm.
  Interventions: Other: Straumann Standard Plus implant and JDental care (JD) Octa implant
- JDental care Octa (JD Octa) (Experimental): Patients receiving JD Octa implants of 4.3 mm in diameter and 10 mm in length.
  Interventions: Other: Straumann Standard Plus implant and JDental care (JD) Octa implant

INTERVENTIONS:
Other: Straumann Standard Plus implant and JDental care (JD) Octa implant — Two different implant systems were used. The above-mentioned implants share many features in common, such as implant design. They both have a machined implant collar of 1.8 mm.
  Other Names: Straumann SP implants; JD Octa implants (J Dental Care)

SUMMARY:
The objective of this prospective study is to compare clinically and radiographically two different tissue-level implants, in partially edentulous patients in the posterior area of the maxilla and mandible. The primary objective of the study was to track the crestal bone level changes around the two implant systems. Secondary objectives were implant stability as well as initial soft tissue thickness which were evaluated throughout this study.

DETAILED DESCRIPTION:
The study is designed as a prospective clinical trial with a parallel design comparing two different tissue-level implants placed adjacently in the posterior maxilla and mandible. The primary outcome is the change in the interproximal crestal bone level.

Patients in this study were recruited from the general population attending the department of Periodontology at the Saint-Joseph University. Adult patients (males and females) in need of implant rehabilitation for partial edentulism in the posterior maxilla and mandible have been selected to take part in this study. Following initial screening procedures, each patient underwent a site-specific intraoral and radiographic examination (Cone Beam Computed Tomography analysis and periapical radiographs) in order to make sure that the inclusion criteria were satisfied. Patients presenting with bone width of less than 6 mm or more than 9 mm were immediately excluded from the study. The day of the surgery, each implantation site was given a number depending on the tooth missing. Then, using a random team generator software each site was randomly assigned to one of the two groups based on the implant system used:

The first group (group 1) consisted of patients receiving Straumann Standard Plus (SP) implants of 4.1 mm in diameter and length of 10 mm.

The second group (group 2) included patients receiving JD Octa implants of 4.3 mm in diameter and 10 mm in length.

Participants were blinded as to the assignment in the first or second group. The implant placement procedures were planned based on clinical and radiographic evaluation.

The following parameters were monitored for each case:

Crestal bone level changes (CBL)

Primary and secondary implant stability

Initial soft tissue thickness

After a healing time of 3 months Patients were recalled 6 and 12 months after prosthetic treatment. At each visit, the restorations were evaluated for mobility, oral hygiene, peri-implant soft tissue conditions and patient satisfaction. Intraoral standardized radiographs were also taken at the 12-months follow-up visit to evaluate crestal bone level changes. CBL changes were defined as the difference between two consecutive CBL measurements. Secondary implant stability was evaluated. Impressions were taken at the implant level. Abutments were fixed on the implants with titanium screws.

In order to reduce the risk of bias in the study, all the implant-supported crowns were screw retained. However, in only one case, and due to prosthetic considerations, two implant-supported crowns were cemented using a temporary cement. In this case, the restorations were thoroughly checked for excessive cement.

Final restorations were delivered within 2 weeks of referral. Finally, standardized radiographs were taken to ensure abutment seating and check for residual cement (in the case of cemented crowns).

Patients were recalled 6 and 12 months after prosthetic treatment. At each visit, the restorations were evaluated for mobility, oral hygiene, peri-implant soft tissue conditions and patient satisfaction. Intraoral standardized radiographs were also taken at the 12-months follow-up visit to evaluate crestal bone level changes. As described previously, CBL changes were defined as the difference between two consecutive CBL measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18, requiring placement of at least two adjacent implants in the posterior maxilla or mandible (premolar-molar area)
* Patients willing to sign the consent form and respect the follow-up period of the study
* Non-smokers or light smokers (less than 10 cig/day)
* No bone augmentation procedures before or during implant placement in the area of interest
* Healthy soft tissue conditions (full mouth plaque scores < 20% and full mouth bleeding index < 20%)
* Minimum height of 2 mm of keratinized tissue
* Minimum of 6 mm in bone width and 10 mm in bone height
* Minimal distance of 2 mm between predicted implant tip and inferior alveolar nerve
* Healed sockets (at least 4 months post-extraction)

Exclusion Criteria:

* Patients not satisfying the inclusion criteria
* Patients with any local or systemic disease
* Patients taking any kind of medication that interferes with bone metabolism
* Pregnant or breast-feeding women
* Patients with parafunctional disorders
* Patients with poor oral hygiene
* Heavy smokers (>10 cig/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Crestal bone level changes. | Radiographic evaluation took place at three time periods: at implant placement, at implant loading and one year after implant loading.
  Peri-implant CBL changes were assessed using periapical radiographs. Radiographs were taken according to the long cone, paralleling technique, using a positioner (XCP Rinn holders, Dentsply Friadent Schweiz, Nidau, Switzerland) parallel to the implant axis and perpendicular to the cone of rays. An individualized radiographic mount (foam and acrylic) was used for each patient to standardize the periapical radiographs. This technique allows the repositioning of the image plate in future radiologic examinations. For the digital process, an image measuring program, Image J (Wayne Rasband, National Institutes of Health) was used.

SECONDARY OUTCOMES:
Initial soft tissue thickness. | Vertical soft tissue thickness was measured immediately during the implant placement.
  Vertical soft tissue thickness was measured with a periodontal probe (PCP-UNC 15; Hu-Friedy, Chicago, IL) placed at the center of the future implant site after full thickness buccal flap elevation.
Primary and secondary implant stability. | Primary and secondary implant stability were measured immediately after implant placement (t1) and after 3 months (t2) respectively.
  Primary and secondary implant stability were measured with Osstell ISQ (Osstell AB, Gothenburg, Sweden).

CONTACTS AND LOCATIONS:
Overall Officials: Carole Chakar, DDS, PhD, Study Director — Head of the department of periodontology
Locations (1):
- Saint Joseph University (USJ), Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Study protocol